CLINICAL TRIAL: NCT06053372
Title: Leveraging Wearable Technologies for Arrhythmia Detection in Children - The PAW (Pediatric Apple Watch) Study
Brief Title: Pediatric Apple Watch Study
Acronym: PAWS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Scott Ceresnak, Professor of Pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 67366
Record Dates: First submitted 2023-09-14; First posted 2023-09-25 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Arrhythmia in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Apple Watch (Experimental): Participants will wear an Apple Watch for 6 months
  Interventions: Device: Apple Watch

INTERVENTIONS:
Device: Apple Watch — Wearable monitor for heart rate and arrhythmia detection

SUMMARY:
Specific Aim #1 - To determine the accuracy of Apple Watch ECG tracings heart rate in children.

Specific Aim #2 - To determine if extended monitoring with the Apple Watch can identify arrhythmia events that were not detected by short term clinical monitoring.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients age 6 - 21 years undergoing clinically indicated arrhythmia monitoring
* Patients with developmental ability (as determined by patient and parents) to safely wear the Apple Watch and utilize the patient activated trigger buttons on both the clinical monitor and the Apple Watch.

Exclusion Criteria:

* Age < 6 years. Those under 6 many not be able to safely use the watch and have the developmental ability (as gauged by clinician and parents) to utilize the trigger features on the watch and cardiac rhythm monitor.
* Inability to effectively utilize the triggered features of the monitor or watch
* Patients unable to utilize the Apple Watch.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Heart rate correlation | Up to 2 weeks
  Comparison of heart rate (bpm) between the Apple Watch and standard clinical rhythm monitor
Arrhythmia correlation | Up to 6 months
  Comparison of the number of clinically significant arrhythmia events between the Apple Watch and standard clinical rhythm monitor. Clinically significant arrhythmia events include supraventricular arrhythmias, ventricular arrhythmias, sinus pauses, and conduction abnormalities/heart block

CONTACTS AND LOCATIONS:
Overall Officials: Scott Ceresnak, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No